CLINICAL TRIAL: NCT01065766
Title: Re-examination Study for General Drug Use to Assess the Safety and Efficacy Profile of JANUMET in Usual Practice
Brief Title: Sitagliptin/Metformin (JANUMET) Re-examination Study (0431A-182)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431A-182; 2010_006 (Other: Merck)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2014-04-17 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Korean participants with type 2 diabetes mellitus treated with sitagliptin/metformin
  Interventions: Drug: Sitagliptin/metformin

INTERVENTIONS:
Drug: Sitagliptin/metformin — Sitagliptin/metformin 50/500 mg, 50/850 mg, or 50/1000 mg tablet administered twice daily with meals.
  Other Names: JANUMET

SUMMARY:
This survey is conducted for preparing application materials for re-examination under the Pharmaceutical Affairs Laws and its Enforcement Regulation, its aim is to reconfirm the clinical usefulness of sitagliptin/metformin (JANUMET) through collecting the safety and efficacy information according to the Re-examination Regulation for New Drugs.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Is treated with sitagliptin/metformin within local label for the first time

Exclusion Criteria:

* Has a contraindication to sitagliptin/metformin according to the local label
* Is treated with sitagliptin/metformin before contract and out of enrollment period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean participants with type 2 diabetes mellitus treated with sitagliptin/metformin in usual practice
Sampling Method: Probability Sample
Enrollment: 4065 (Actual)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this post-marketing surveillance study of sitagliptin/metformin (JANUMET®), participants in South Korea treated for >= 24 weeks were evaluated for long-term safety and efficacy. During the re-examination study period (December 4, 2005 to September 20, 2013), case report forms (CRFs) were collected from 4,065 participants.
Groups:
- All Participants Included in the Safety Evaluation: Korean participants with type 2 diabetes mellitus treated with sitagliptin/metformin
Period: Overall Study
Arm/Group | All Participants Included in the Safety Evaluation
Started | 4065
Completed | 4033
Not Completed | 32
Not completed — Assessed before the contracted date | 1
Not completed — Contraindication to administration | 6
Not completed — Violated dosage/administration | 25

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only reported for the Safety Population (4033) who qualified for the study and not for the 4065 participants from whom CRFs were collected.
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 4033
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.22 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1913
  Male | 2120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Experience
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 26 weeks
Population: All participants who were included in the safety evaluation
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 4033
Percentage of participants | 3.74

2. Primary Outcome: Change From Baseline to Treatment in Hemoglobin HbA1c (A1C) at Week 12
Description: HbA1C is found when high blood levels of glucose combines with hemoglobin to form glycated hemoglobin. The average amount of glucose in blood over a prolonged periods of time can be determined by measuring a hemoglobin A1c level which is reported as a percentage (%). The change from baseline reflects the Week 12 A1C minus Week 0 A1C.
Time Frame: Baseline and Week 12
Population: All participants with a pre-treatment and a 12-week post-treatment HbA1c value.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 1597
Percentage of glycosylated hemoglobin | -0.93 (1.23)

3. Primary Outcome: Change From Baseline to Treatment in Fasting Plasma Glucose (FPG) at Week 12
Description: Blood glucose was measured on a fasting basis (collected after an 8- to 10-hour fast). FPG is expressed as mg/dL. Therefore, this change from baseline reflects the Week 12 FPG minus Week 0 FPG.
Time Frame: Baseline and Week 12
Population: Participants with a pre-treatment and a 12-week post-treatment measurement of FPG.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 1343
mg/dL | -28.21 (42.21)

4. Primary Outcome: Change From Baseline in 2-hour Post Prandial Glucose (2hr-PPG) at Week 12
Description: Blood glucose was measured 2 hours after a meal (2hr-PPG). 2hr-PPG is expressed as mg/dL. Therefore, this change from baseline reflects the Week 12 2hr-PPG minus Week 0 2hr-PPG.
Time Frame: Baseline and Week 12
Population: Participants with a pre-treatment and a 12-week post-treatment measurement of 2hr-PPG.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 1219
mg/dL | -58.02 (72.96)

5. Primary Outcome: Percentage of Participants With an Overall Efficacy Evaluation by the Investigator of Improved, Stable, or Worse at Week 12
Description: Overall efficacy analysis was conducted on participants who have used study drug for more than 12 weeks and whose improvement of the disease has been assessed by Principal investigator. The investigator's global assessment of disease improvement was classified as either: "Improved", "Stable" and "Worse" in a Medical History/Physical Examination form.
Time Frame: At Week 12
Population: Participants who have used study drug for more than 12 weeks and whose improvement of the disease has been assessed by Principal investigator.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 3241
Percentage of participants
  Improved | 78.68
  Stable | 16.38
  Worse | 4.94

6. Primary Outcome: Change From Baseline to Treatment in HbA1c at Week 24
Description: HbA1C is blood marker used to report average blood glucose levels over a prolonged periods of time and is reported as a percentage (%). Therefore, this change from baseline reflects the Week 24 A1C minus Week 0 A1C.
Time Frame: Baseline and Week 24
Population: All participants with a pre-treatment and a 24-week post-treatment HbA1c value.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated hemoglobin
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 347
Percentage of glycosylated hemoglobin | -1.08 (1.42)

7. Primary Outcome: Change From Baseline to Treatment in FPG at Week 24
Description: Blood glucose was measured on a fasting basis (collected after an 8- to 10-hour fast). FPG is expressed as mg/dL. Therefore, this change from baseline reflects the Week 24 FPG minus Week 0 FPG.
Time Frame: Baseline and Week 24
Population: Participants with a pre-treatment and a 24-week post-treatment measurement of FPG.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 230
mg/dL | -32.40 (44.75)

8. Primary Outcome: Change From Baseline in 2hr-PPG at Week 24
Description: Blood glucose was measured 2 hours after a meal (2hr-PPG). 2hr-PPG is expressed as mg/dL. Therefore, this change from baseline reflects the Week 24 2hr-PPG minus Week 0 2hr-PPG.
Time Frame: Baseline and Week 24
Population: Participants with a pre-treatment and a 24-week post-treatment measurement of 2hr-PPG.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 218
mg/dL | -62.13 (75.67)

9. Primary Outcome: Percentage of Participants With an Overall Efficacy Evaluation by the Investigator of Improved, Stable, or Worse at Week 24
Description: Overall efficacy analysis was conducted on participants who have used study drug for more than 24 weeks and whose improvement of the disease has been assessed by Principal investigator. The investigator's global assessment of disease improvement was classified as either: "Improved", "Stable" and "Worse" in a Medical History/Physical Examination form.
Time Frame: At Week 24
Population: Participants who have used study drug for more than 24 weeks and whose improvement of the disease has been assessed by Principal investigator.
Measure: Number; unit: Percentage of participants
Arm/Group | All Participants Included in the Safety Evaluation
Number analyzed (Participants) | 800
Percentage of participants
  Improved | 76.38
  Stable | 15.88
  Worse | 7.75

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Arm/Group | All Participants Included in the Safety Evaluation
Serious Adverse Events (participants affected / at risk) | 17/4033
Other Adverse Events (participants affected / at risk) | 0/4033
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Included in the Safety Evaluation (N=4033)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
CHRONIC HEPATITIS C (Infections and infestations) | 1 (2)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
THYROID NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
TENSION HEADACHE (Nervous system disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
KNEE ARTHROPLASTY (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In regard to surveillance result, any publication should be agreed by sponsor in advance.